CLINICAL TRIAL: NCT01168908
Title: Phase 2 Clinical Trial of Sildenafil for Cardiac Dysfunction in Duchenne Muscular Dystrophy and Becker Muscular Dystrophy
Brief Title: Revatio for Heart Disease in Duchenne Muscular Dystrophy and Becker Muscular Dystrophy
Acronym: REVERSE-DBMD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: As recommended by the DSMB.
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Kathryn Wagner, Associate Professor of Neurology, Johns Hopkins University School of Medicine, Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NA-00036602
Record Dates: First submitted 2010-07-22; First posted 2010-07-23 (Estimated); Results first posted 2018-03-21 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Duchenne Muscular Dystrophy; Becker Muscular Dystrophy
Keywords: Clinical trial; Revatio; Sildenafil; Muscular Dystrophy; Duchenne; Becker; Adult; Adolescent
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophies | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Revatio (sildenafil) (Experimental): This arm will receive Revatio (sildenafil) for 12 months. During the first 6 months, the subject and investigator will be blinded to treatment. The second 6 months, will be open label treatment with Revatio.
  Interventions: Drug: Sildenafil
- Placebo (Other): This arm will receive placebo (sugar pill) for 6 months and Revatio (sildenafil) for 6 months. During the first 6 months, the subject and investigator will be blinded to treatment. The second 6 months, will be open label treatment with Revatio.
  Interventions: Drug: Sildenafil

INTERVENTIONS:
Drug: Sildenafil — 20mg tablet three times daily
  Other Names: Revatio

SUMMARY:
This study, supported by Charley's Fund, Inc., is being done to determine if the drug Revatio®(also known as Sildenafil), as compared to placebo (an inactive substance that looks like the study drug, but contains no medication), improves heart function in people with Duchenne Muscular Dystrophy and Becker Muscular Dystrophy (DBMD).

In people with DBMD, dystrophin is not present or lacking in heart and muscle. This is associated with abnormalities in an enzyme called "neuronal nitric oxide synthase" or nNOS, and leads to decreases in "cyclic GMP," which is necessary for proper function of those muscles. Revatio blocks an enzyme called phosphodiesterase 5 (PDE5), and helps to restore the normal amounts of cyclic GMP. The purpose of this research is to determine if Revatio is safe for people with DBMD and if it can improve heart function.

Hypothesis : PDE5 inhibition, with the use of Revatio, will improve cardiac function in patients with DBMD.

DETAILED DESCRIPTION:
This clinical trial is focused on cardiovascular disease due to dystrophin deficiency. Dystrophin is normally localized to the muscle cell membrane where it interacts with a complex of proteins including neuronal nitric oxide synthase (nNOS). DMD gene mutations lead to the loss of dystrophin and to mislocalization and reduced activity of nNOS, consequently reducing cyclic guanosine monophosphate (cGMP) and the activity of its downstream effector, protein kinase G. Our group and others have shown that inhibition of phosphodiesterase 5 (PDE5) leads to favorable cardiac remodeling and improved vascular tone in animal models of heart failure.

This will be a phase 2, randomized, double-blind, placebo-controlled single center study for 6 months followed by open-label period of 6 months in which all enrolled subjects receive Revatio (a PDE5 inhibitor). A single dose of Revatio (20 mg three times daily) will be tested based on the safety and efficacy of that dose for treatment of pulmonary hypertension.

The primary endpoint will be the change in cardiac left ventricular end-systolic volume (LVESV) as determined by cardiac MRI after 6 months of Revatio compared to baseline. A 10% change in LVESV will be considered significant. This degree of improvement has generally been observed in cardiac therapies that improve survival such as ACE inhibitors, beta blockers, and cardiac resynchronization. The change from baseline in LVESV after 6 months of Revatio will be compared to the change in LVESV over 6 months with placebo. The study will extend for an additional 6 months of open-label Revatio to provide data on 6 months versus 12 months of Revatio treatment. Additional secondary endpoints will include differences in systolic and diastolic LV function by MRI, differences in LV mass and fibrosis by MRI, brachial flow-mediated vasodilation (peripheral endothelial function), and targeted exploratory assessment of differences in skeletal muscle function using forced vital capacity (FVC) and pincher and grip testing. Safety will be assessed by differences in the frequency and grade of adverse events

The study is taking place at the Kennedy Krieger Institute/Johns Hopkins Medical Institutions in Baltimore, MD. The trial requires out-patient visits over a 12-month period. Travel funds, through a grant from Ryan's Quest, are available.

ELIGIBILITY:
Inclusion Criteria:

1. DBMD as determined by either a skeletal muscle biopsy demonstrating absence or lack of dystrophin, and/or genetic testing showing a mutation in the dystrophin gene predictive of DBMD, as well as a consistent physical examination
2. Male gender
3. Age greater than or equal to 18 years
4. Cardiac dysfunction with ejection fraction less than or equal to 50% as determined by echocardiogram, cardiac MRI, or multi-gated acquisition (MUGA) scan
5. On a stable dose of ACE-inhibitor or angiotensin receptor blocker (ARB) for at least 3 months; beta-adrenergic receptor blockers and glucocorticosteroids are not required but if used, a stable dose for at least 3 months is required.
6. Ability of the subject or legal guardian to provide informed consent
7. Ability to adhere with study follow-up
8. Willingness to abstain from food and alcohol for 8 hours prior to FMD

Exclusion Criteria:

1. Use of nitrates or alpha-adrenergic receptor blockers
2. Known intolerance or allergy to sildenafil, or a history of any severe allergic or anaphylactic reactions
3. Any medical or psychosocial condition, which, in the view of the study investigator, makes study participation inadvisable
4. Known hereditary retinal disorder such as retinitis pigmentosa
5. History of priapism or conditions that may predispose to priapism such as sickle cell anemia, multiple myeloma, or leukemia
6. Bleeding disorders
7. Active tobacco use
8. Chronic atrial fibrillation or frequent arrhythmia that would result in an irregular pulse
9. Factors that would preclude obtaining an MRI study - (e.g. implantable pacemaker or cardioverter-defibrillator; body habitus cannot fit into scanner)
10. Systolic blood pressure (SBP) less than 85 mmHg at baseline evaluation
11. Chronic kidney disease stages 4 and 5: GFR< 30 mL/min/1.73 m2 as determined by serum cystatin C level and the equation eGFRcys = 76.7 x (serum cystatin C-1.18)
12. Current use of sildenafil.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-09; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel P Judge, MD, Principal Investigator — Johns Hopkins School of Medicine; Kathryn R. Wagner, M.D., Ph.D., Principal Investigator — The Kennedy Krieger Institute
Locations (1):
- Kennedy Krieger Institute, Johns Hopkins School of Medicine, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Leung DG, Herzka DA, Thompson WR, He B, Bibat G, Tennekoon G, Russell SD, Schuleri KH, Lardo AC, Kass DA, Thompson RE, Judge DP, Wagner KR. Sildenafil does not improve cardiomyopathy in Duchenne/Becker muscular dystrophy. Ann Neurol. 2014 Oct;76(4):541-9. doi: 10.1002/ana.24214. Epub 2014 Jul 10. PMID 25042693

RESULTS

PARTICIPANT FLOW:
Period: Double Blind, Placebo Controlled
Arm/Group | Revatio (Sildenafil) | Placebo
Started | 10 | 10
Completed | 7 | 8
Not Completed | 3 | 2
Period: Open Label
Arm/Group | Revatio (Sildenafil) | Placebo
Started | 7 | 8
Completed | 6 | 7
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Revatio (Sildenafil) | Placebo | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.5 (8.2) | 22.6 (4.4) | 24.05 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 10 | 10 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 7 | 8 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Cardiac Left Ventricular End-systolic Volume (LVESV) by Cardiac Magnetic Resonance (CMR) Imaging.
Description: To determine whether a 6 month trial of oral sildenafil compared to placebo improves cardiac contractile function in DBMD as determined by a > 10% decline in end-systolic volume as detected by CMR.
Time Frame: 6 months compared to baseline
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Revatio (Sildenafil) | Placebo
Number analyzed (Participants) | 7 | 8
ml | 5.2 (23.61) | -0.19 (5.56)

2. Secondary Outcome: Change in Cardiac Systolic and Diastolic Function by CMR
Description: Cardiac volumes and systolic ejection parameters will be measured.
Time Frame: 6 months and 12 months
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Revatio (Sildenafil) | Placebo
Number analyzed (Participants) | 7 | 8
ml
  LV end-diastolic volume | 5.54 (18.85) | 0.24 (8.78)
  stroke volume | 0.34 (9.75) | 0.43 (11.46)

3. Secondary Outcome: Change in Cardiac Mass
Description: Left ventricular (LV) mass will be measured by CMR .
Time Frame: 6 months and 12 months
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Revatio (Sildenafil) | Placebo
Number analyzed (Participants) | 7 | 8
grams | -3.4 (7.03) | -1.05 (12.69)

4. Secondary Outcome: Change in Forced Vital Capacity (FVC) by Pulmonary Function Testing
Description: Skeletal muscle function of the diaphragm will be measured using FVC by pulmonary function testing.
Time Frame: 6 months and 12 months
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Revatio (Sildenafil) | Placebo
Number analyzed (Participants) | 7 | 8
liters | -0.13 (0.09) | -0.19 (0.21)

5. Secondary Outcome: Change in Skeletal Muscle Strength
Description: Skeletal muscle strength will be assessed by pincher and grip dynamometry
Time Frame: 6 months and 12 months
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Revatio (Sildenafil) | Placebo
Number analyzed (Participants) | 7 | 8
pounds
  pinch strength | -0.06 (0.30) | 0.12 (0.45)
  grip strength | 0.37 (0.90) | 0.17 (1.25)

6. Secondary Outcome: Ejection Fraction
Description: Left ventricular ejection fraction by cardiac MRI was measured
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percentage of volume
Arm/Group | Revatio (Sildenafil) | Placebo
Number analyzed (Participants) | 7 | 8
percentage of volume | 43.25 (12.82) | 45.64 (6.82)

ADVERSE EVENTS:
Arm/Group | Revatio (Sildenafil) | Placebo
All-Cause Mortality (participants affected / at risk) | 1/18 | 0/10
Serious Adverse Events (participants affected / at risk) | 5/18 | 1/10
Other Adverse Events (participants affected / at risk) | 13/18 | 7/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Revatio (Sildenafil) (N=18) | Placebo (N=10)
Death from heart failure (Cardiac disorders) | 1 (1) | 0 (0)
dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Prostate infection (Infections and infestations) | 1 (1) | 0 (0)
fecal impaction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Revatio (Sildenafil) (N=18) | Placebo (N=10)
Dizziness (General disorders) | 1 (1) | 0 (0)
gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
low blood pressure (Cardiac disorders) | 4 (4) | 0 (0)
flushing (General disorders) | 1 (1) | 1 (1)
gastroenteritis (Gastrointestinal disorders) | 2 (2) | 1 (1)
tingling sensation (General disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No